CLINICAL TRIAL: NCT01719640
Title: Autologous Bone Marrow Mesenchymal Stem Cell and Bone Marrow Mononuclear Cell Infusion in Type 2 Diabetes Mellitus
Brief Title: MSC and MC in Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fuzhou General Hospital (Other)
Responsible Party: Principal Investigator, Jianming Tan, Professor, Fuzhou General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MSC-MC-DM
Record Dates: First submitted 2012-10-06; First posted 2012-11-01 (Estimated); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: mesenchymal stem cells; bone marrow mononeclear cells; type 2 diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MSC+MC (Experimental): infusion of BMMSC+BMMNC and insulin injection
  Interventions: Drug: infusion of MSCs; Drug: infusion MCs; Drug: insulin
- MC (Active Comparator): infusion of BMMNC and insulin injection
  Interventions: Drug: infusion MCs; Drug: insulin
- Insulin (Active Comparator): insulin injection
  Interventions: Drug: insulin

INTERVENTIONS:
Drug: infusion of MSCs — infusion of MSCs
  Arms: MSC+MC
Drug: infusion MCs — infusion of MCs
  Arms: MC; MSC+MC
Drug: insulin — intensive insulin care

SUMMARY:
Cell injury in human islets induced by non-immune mediated inflammation occur in vitro upon hyperglycemia in type 2 diabetes mellitus. Infusion of autologous bone marrow mononuclear cells (MCs) is an emerging therapeutic approach for DM, which showed promising outcomes with mild side effects. Infusion of MCs and autologous bone marrow mesenchymal stem cells in combination might exert enhanced repairing effects. We hypothesized that infusion of these two classes of cells might provide multiple signals for regeneration and improve recovery from inflammation-induced lesion. The effects might be maximized by intra-arterial pancreatic infusion.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent.
* Mentally stable and able to comply with the procedures of the study protocol.
* Clinical history compatible with type 2 diabetes (T2DM) as defined by the Expert Committee on the Diagnosis and classification of Diabetes Mellitus
* Onset of T2DM disease at ≥ 35 years of age.
* T2DM duration ≥ 3 and ≤ 20 years at the time of enrollment.
* Basal C-peptide 0.3-2.0 ng/mL
* HbA1c ≥ 7.5 and ≤ 12% before standard medical therapy (SMT). Patients must have been treated with SMT for minimum of 4 months prior to randomization.

Insulin dose and metformin doses should be stable over the 3 months prior to randomization.

* HbA1c ≥ 7.5 and ≤ 9.5% at time of randomization.
* Total insulin daily dose (TDD) at time of randomization should not exceed 1.0 units/day/kg

Exclusion Criteria:

* BMI >35 kg/m2.
* Insulin requirements of > 100 U/day.
* HbA1c >9.5%. (at the time of randomization)
* C-reactive protein (hs-CRP) >3.00
* Uncontrolled blood Pressure: SBP >160 mmHg or DBP >100 mmHg at the time of randomization.
* Evidence of renal dysfunction, serum creatinine > 1.5 mg/dl (males) and 1.4 mg/dl (females).
* Proteinuria > 300 mg/day
* Evidence of cardiovascular disease, existing congestive cardiac failure on physical exam and/or acute coronary syndrome in past 6 months.
* For female participants: Positive pregnancy test, presently breast-feeding, or unwillingness to use effective contraceptive measures for the duration of the study.For male participants: intent to procreate 3 months before or after the intervention or unwillingness to use effective measures of contraception. Oral contraceptives,Norplant®, Depo-Provera®, and barrier devices with spermicide are acceptable contraceptive methods; condoms used alone are not acceptable
* Active infection including hepatitis C, HIV, or TB as determined by a positive skin test or clinical presentation, or under treatment for suspected TB. Positive tests are acceptable only if associated with a history of previous vaccination in the absence of any sign of active infection. Positive tests are otherwise not acceptable, even in the absence of any active infection at the time of evaluation
* Known active alcohol or substance abuse including cigarette/cigar smoking
* Baseline Hgb below the lower limits of normal at the local laboratory; lymphopenia (<1,000/L), neutropenia (<1,500/L), or thrombocytopenia (platelets <100,000/L).
* A history of Factor V deficiency or other coagulopathy defined by INR >1.5, PTT>40, PT >15.
* Any coagulopathy or medical condition requiring long-term anticoagulant therapy(e.g., warfarin) after transplantation (low-dose aspirin treatment is allowed) or patients with an INR >1.5.
* Acute or chronic pancreatitis.
* Symptomatic peptic ulcer disease.
* Hyperlipidemia despite medical therapy (fasting LDL cholesterol >130 mg/dl, treated or untreated; and/or fasting triglycerides > 200 mg/dl).
* Receiving treatment for a medical condition requiring chronic use of systemic steroids.
* Symptomatic cholecystolithiasis.
* Use of any investigational agents within 4 weeks of enrollment.
* Admission to hospital for any reason in the 14 days prior to enrollment (signing consent).
* Presence of active proliferative diabetic retinopathy or macular edema
* Any malignancy
* Abnormal liver function >1.5 x ULN
* Abdominal aortic aneurysm
* History of cerebro-vascular accident
* Any patient with acute or subacute decompensation from diabetes
* Any acute or chronic infectious condition that in the criteria of the investigator would be a risk for the patient.
* Subjects with hypoproteinemia, cachexia or terminal states
* Subjects with history of anorexia/bulimia
* Subjects with respiratory insufficiency
* Subjects that are being treated with any medication that could interfere with the outcome of the study such as: Sulfonylureas, Thiazolidinediones and glucagon like peptide 1 (GLP-1) analogues (Exenatide, Byetta), Pramlintide (Amylin), Dipeptidylpeptidase IV (DPP-IV) inhibitors (i.e. Sitagliptin, Januvia)
* Any medical condition that, in the opinion of the investigator, will interfere with thesafe completion of the trial.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2013-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
macrovascular complications | 8 years
microvascular complications | 8 years

SECONDARY OUTCOMES:
DPN | 8 years
  diabetes peripheral neuropathy
MI | 8 years
  myocardial infarction
angina | 8 years
  angina
stroke | 8 years
  stroke
amputation | 8 years
  amputation
DN | 8 years
  diabetes nephropathy
DRP | 8 years
  diabetes retinopathy
pro-DRP | 8 years
  proliferative diabetes retinopathy
C-peptide AUC | 1y
  C-peptide area under the curve
insulin AUC | 1y
  insulin area under the curve
HbA1c | 1y
  glycated hemoglobin
FBG | 1y
  fasting hemoglucose
insuline dose | 1y
  exogenous insulin requirements
fasting C-p | 1y
  fasting c-peptide
The incidence and severity of adverse events related to the stem cell infusion procedure | 8y

CONTACTS AND LOCATIONS:
Locations (1):
- Fuzhou General Hospital, Xiamen Univ, Fuzhou, Fujian, China

REFERENCES:
- [Derived] Wu Z, Huang S, Li S, Cai J, Huang L, Wu W, Chen J, Tan J. Bone marrow mesenchymal stem cell and mononuclear cell combination therapy in patients with type 2 diabetes mellitus: a randomized controlled study with 8-year follow-up. Stem Cell Res Ther. 2024 Sep 30;15(1):339. doi: 10.1186/s13287-024-03907-w. PMID 39350270